CLINICAL TRIAL: NCT00792844
Title: Comparison of Two Formulations of Lactobacillus Acidophilus and Lactobacillus Casei in the Prevention of Antibiotic-Associated Diarrhea: a Pilot Study
Brief Title: Comparison of Two Formulations of Bio-K
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Gloria Seto, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-Seto
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2008-11-18 (Estimated); Status verified 2008-11

CONDITIONS: Antibiotic-Associated Diarrhea
MeSH Terms: interventions — Dosage Forms

ARMS (3):
- Bio-K capsule (Experimental): 1 capsule of lactobacillus acidophilus and lactobacillus casei (50 billion live bacteria) daily for duration of antibiotic therapy and 7 days after or until discharge, whichever comes first
  Interventions: Dietary Supplement: Bio-K capsule formulation
- Bio-K liquid (Active Comparator): 98 g of lactobacillus acidophilus and lactobacillus casei (50 billion live bacteria) daily for the duration of antibiotic treatment and for 7 days after termination of antibiotics or until hospital discharge, whichever comes first
  Interventions: Dietary Supplement: Bio-K drink
- no Bio-K (No Intervention): No lactobacillus product - standard infection control procedures (i.e. handwashing, etc.)

INTERVENTIONS:
Dietary Supplement: Bio-K capsule formulation — Bio-K 1 capsule formulation daily for the duration of antibiotic treatment and for 7 days after termination of antibiotics or until hospital discharge, whichever occurs first
  Arms: Bio-K capsule
Dietary Supplement: Bio-K drink — Bio-K 98 g of diary-free soy beverage formulation for the duration of antibiotic treatment and for 7 days after termination of antibiotics or until hospital discharge, whichever occurs first
  Arms: Bio-K liquid

SUMMARY:
Main research Question: The investigators would like to find out if both the Bio-K (lactobacillus acidophilus and lactobacillus casei) drink and capsule are equally effective in the prevention of diarrhea associated with antibiotic use.

Why is this research project important? About 25% of patients who use antibiotics may develop diarrhea as a side effect. Symptoms are mild and consist of watery diarrhea and abdominal pain. Some patients may develop a more severe form of diarrhea, called clostridium difficile-associated diarrhea. Clostridium difficile-associated diarrhea may lead to more serious consequences like inflammation of the large bowel and in some cases, death. There are some studies that suggest Bio-K drink, a probiotic preparation containing lactobacillus acidophilus and lactobacillus casei, decreases the risk of diarrhea from antibiotic use. As a result, St. Joseph's Healthcare has recently to use Bio-K routinely to try to reduce risk of patients developing diarrhea. No other Hamilton hospitals use Bio-K routinely as there is not strong evidence about the effectiveness of Bio-K for the prevention of diarrhea. This study will provide more information about Bio-K's effectiveness in the prevention of diarrhea associated with antibiotic use as both a capsule and a drink.

ELIGIBILITY:
Inclusion Criteria:

* speak English
* capable of providing consent
* reachable by telephone within the next three months
* willing to comply with study protocols
* age over 65 years
* prescribed clindamycin, fluoroquinolones or cephalosporin for more than one dose

Exclusion Criteria:

* ICU patients
* transplant patients
* patients on immunosuppressant medications (prednisone greater than 50 mg/day for 7 days, azathioprine, cyclosporine, cyclophosphamide, tacrolimus, sirolimus, methotrexate, mycophenolate, anti-TNF agents, interleukin-2 chemotherapy)
* HIV patients with CD4+ count less than 250 cells/mm3
* neutropenic patients with total neutrophil count less than 500
* patients with prosthetic heart valves

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-02; Primary Completion 2009-05 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Antibiotic-associated diarrhea | 30 days after termination of antibiotic

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton - Charlton Campus, Hamilton, Ontario, Canada